CLINICAL TRIAL: NCT03855735
Title: "Sufficiency, Accuracy, Clarity, Contextualization, and Interpersonal Adaptation - Safe, Digitally Supported Communication in Gynecology and Obstetrics: TeamBaby"
Brief Title: TeamBaby - Safe, Digitally Supported Communication in Obstetrics and Gynecology
Acronym: TeamBaby
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobs University Bremen gGmbH (Other)
Collaborators: German Coalition for Patient Safety (Aktionsbündnis Patientensicherheit) (Unknown); Techniker Krankenkasse (Other); University Hospital Ulm (Other); The German Innovation Fund (Innovationsfonds) (Unknown); Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Sonia Lippke, Principal Investigator and Professor of Health Psychology & Behavioral Medicine, Jacobs University Bremen gGmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCT03855735; 01VSF18023 (Other Grant/Funding Number: The Federal Joint Committee (G-BA))
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy Related
Keywords: Preventable adverse events; Patient safety; Core communication competences; Different communication models; HAPA; Participatory intervention development; Digitization; App; eHealth; Health services research
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Parallel design for Phase 2 and sequential design in Phase 3
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TeamBaby Online Training Intervention Group Phase 2 (IG1) (Experimental): Those who give birth and relatives who have been arbitrarily assigned to the intervention group receive an interactive online training on different communication models and competencies (Phase 2).
  Interventions: Behavioral: TeamBaby Online Communication Training (IG1) and TeamBaby Web-App Communication Training (IG2)
- No Intervention (No Intervention): Those who give birth and relatives who have been arbitrarily assigned to the control group do not receive any training on different communication models competencies and will not gain access to the digital app prior to giving birth.
- TeamBaby App Training Intervention Group Phase 3 (IG2) (Experimental): Those who give birth and relatives who have been arbitrarily assigned to the intervention group will gain access to the digital app and receive a communication training via the app (Phase 3).
  Interventions: Behavioral: TeamBaby Online Communication Training (IG1) and TeamBaby Web-App Communication Training (IG2)

INTERVENTIONS:
Behavioral: TeamBaby Online Communication Training (IG1) and TeamBaby Web-App Communication Training (IG2) — The developed short manual for the teaching of different communication models competences will enable those who have been arbitrarily assigned to the intervention group and their relatives to develop secure communication competences (Phase 2). In Phase 3, the intervention group will have access to the digital app.
  Arms: TeamBaby App Training Intervention Group Phase 3 (IG2); TeamBaby Online Training Intervention Group Phase 2 (IG1)

SUMMARY:
The purpose of this project with obstetric healthcare workers, pregnant women and their relatives is to improve communication between all parties involved in order to increase sustainable patient safety. To this end, clinical staff, expectant mothers and their partners as well as relatives will be trained in personal sessions and through digital interventions. The aim is to improve their ability to communicate more confidently with each other. In addition, an app will be developed to support all participants in their communication with each other and in overcoming difficulties in everyday hospital life. The project contributes to reduce the frequency of preventable adverse events (pAEs) in gynecology and obstetrics and to increase patients' satisfaction with their treatment. Data will be collected in three study phases:

1. Implementation phase - Training for obstetric healthcare workers at two German university hospitals which will be developed and implemented based on observations, interviews, and focus groups and pre-experimental study with pre/post-test (questionnaires for participants, interviews). To evaluate patient safety, an analysis of hospital data will be conducted incl. retrospective cohort study;
2. Effectiveness study with randomized controlled study design (questionnaires and interviews). In the intervention group, pregnant women and their relatives will be trained in safe communication;
3. Implementation of an app (evaluated via questionnaires, observations, interviews, focus groups). Women who receive the training via the app will be compared to the historical control group as case-control study (questionnaires, interviews, analysis of hospital data).

DETAILED DESCRIPTION:
Phase 1:

The concept of the needs assessment is based on a previous approach, which aimed to implement an intervention to increase the safety of patient transfers in intensive care units. This should lead to a comprehensive understanding of the beneficial and inhibitory conditions as well as potentials for the implementation of the intervention in the field (e.g., how different communication techniques can be integrated beyond training into clinical practice). Observations for the ethnographic analyses are recorded in a standardized observation protocol. Focus groups and interviews are conducted with partially standardized guidelines with at least one person from each occupational group in order to gain as comprehensive an impression as possible of possible resources and barriers for the implementation of the intervention. The data will then be analyzed in terms of content using an inductive approach and used to develop the training. Migration background will be considered exploratively in the data collection and testing as well as participatory in the app development (i.e. it will be ensured that patients and accompanying persons with migration background will also be included in the development). Different communication models competencies and tailoring based on the Health Action Process Approach (HAPA) will also be integrated into the training and app intervention. A short manual for practical support and written documentation of the training process will be prepared, also to avoid failure of implementation. The online training will be offered in the pre-experimental study to all professionals at both intervention sites. The aim is to investigate the connection between the staff trainings and preventable Adverse Events (pAEs) that are compared between the year 2018 (before the staff trainings) and 2020 (after the staff trainings), to observe mechanisms of action and to create a basis for the implementation of phase 2.

Additional remark 23/06/22: The paper comparing pAEs between 2018 and 2020 is currently under review.

The study regarding the questionnaire evaluation has a one-group, pre-/post-design. The study includes all specialists (e.g. doctors, nurses, midwives, obstetricians) at both locations with a total of N = 140 participants. Specialists are trained in interdisciplinary groups of 10 to 12 participants.

Additional remark 23/06/22: The paper concerning the evaluation of communication behavior and behavioral factors associated with this behavior has been published.

Summary of the implementation phase: Research questions, methods, study population and target criteria

A: What is the prevalence of pAEs? This question will be answered using monitoring protocols and anonymous routine data of the hospital from 2018 in a Mixed Methods study: Quality indicators include the reporting according to safe communication, pAEs, and a retrospective cost analysis of pAEs.

Additional remark 23/06/22: The paper for the evaluation of pAEs has been published.

B: What are effective interventions to optimize communication in everyday hospital life? This question will be answered by updating the status of the literature search in Pubmed, PsychInfo, Cochrane Database to provide an overview of effective interventions and effect strengths.

Additional remark 23/06/22: The systematic review has been published.

C: What is the adherence for equivalent patient safety measures (e.g. hand hygiene)? Using questionnaire data of all employees at both intervention sites to measure adherence to patient safety measures and identify relationships between adherence and quality indicators Additional remark 23/06/22: The paper including questionnaire and observational data has been published.

D: What are possible resources and barriers for the implementation of an intervention in order to optimize communication in everyday hospital life? The question will be answered in Ethnographic observation and guideline-based individual and focus group interviews with physicians, nursing staff, training assistants, psychologists, and midwives to classify resources and barriers.

Additional remark 23/06/22: The according publication has been finalized.

E: What is an appropriate strategy to implement effective interventions to optimize communication? For this question, there will be a triangulation of results from previous steps including the matching of data from interviews, focus groups and questionnaires with evidence from the literature to determine the implementation strategy regarding resources and barriers in implementing the intervention to patient safety.

Additional remark 23/06/22: The triangulation was published.

Since the aim is to achieve full inclusion of all healthcare workers in Phase 1, no inclusion and exclusion criteria are defined. Differences between the measurement times are checked using linear and general mixed models, initial values of the first measurement are taken into account as covariates. Clinics are modeled as a fixed effect. For the entire analysis, corresponding confidence intervals of 95 % are determined. To calculate the standardized mean difference (SMD) between the two measurement points, the non-standardized regression coefficients are standardized to the pooled standard deviation of the observed measured values. According to Cohen's recommendations, SMDs are interpreted as follows: small effect by SMD = 0.2; medium effect by SMD = 0.5; large effect by SMD = 0.8. The odds ratio of binary outcomes is subjected to a logit transformation to calculate effect strengths. To check whether the intervention effect on the primary target criterion is moderated by external variables, reciprocal interaction terms are considered in the model estimation. Continuous moderators are standardized by z-transformation. The estimated parameter of the interaction between the z-transformed continuous variable and the effect estimator of the group difference thus represents the additional intervention effect if the potential moderator increases by a standard deviation. Participants are only included in the analysis if they participate in the corresponding follow-up online survey and are analyzed according to intention to treat. Differences are interpreted as significant when the p-value of a two-sided test is <0.05.

Additional remark 22/06/22: The evaluation of questionnaire data has been published.

Due to the COVID-19 pandemic, the trainings for staff members had to be paused. Although all staff members (N=141) were trained, only N=67 provided questionnaire data at both time points (before and after the training). Hence, the analysis was performed as a MANOVA to evaluate the questionnaire data.

The manuscript evaluating clinical data (preventable adverse events) is currently under review.

Phase 2:

In Phase 2, the effectiveness of the communication intervention for the target group of women giving birth/family members is assessed using the gold standard, i.e. randomized control trial (RCT). In each institution, four employees are enabled to train patients and their relatives on the short manual developed to teach different communication models competencies. When a woman gives birth and her relatives are admitted, they are randomly assigned to a training group (IG) or a control group (CG). The pAEs are collected on a person-specific basis (anonymized) and coded in parallel. With an alpha error of 0.05 and a power of 80%, a sample of N = 352 is necessary (to be analyzed IG: N = 176; CG: N = 176) in order to be able to prove an effect of d = 0.3. With an assumed drop-out of 20%, N = 424 participants (to be recruited IG: N = 212; CG: N = 212) would have to be recruited (recruitment sample). The target criteria are evaluated statistically and clinically as in phase 1. Group differences are checked by means of linear and general mixed models, initial values of the first measurement point are considered as covariates. Clinics are modelled as fixed effects. For the entire analysis, corresponding confidence intervals of 95 % are determined. To calculate the standardized mean difference (SMD) between the two measurement points, the non-standardized regression coefficients are standardized to the pooled standard deviation of the observed measured values. According to Cohen's recommendations, SMDs are interpreted as follows: small effect by SMD = 0.2; medium effect by SMD = 0.5; large effect by SMD = 0.8. The odds ratio of binary outcomes is subjected to a logit transformation to calculate effect strengths. To check whether the primary target criterion is moderated by external variables, reciprocal interaction terms are considered in the model estimation. Continuous moderators are standardized by z-transformation. The estimated parameter of the interaction between the z-transformed continuous variable and the effect estimator of the group difference thus represents the additional intervention effect if the potential moderator increases by one standard deviation. Participants are only included in the analysis if they participate in the corresponding follow-up online survey and are analyzed according to intention to treat. Differences are interpreted as significant when the p-value of a two-sided test is <0.05.

Additional remark 28/06/22: The manuscript regarding the questionnaire data is currently under review. Due to a higher drop-out than originally calculated, the analysis was changed from an ANCOVA to a multilevel linear model to evaluate training effects.

Phase 3:

From all findings in phases 1 and 2, the digital app will be developed in a participatory and theory-driven way. The aim is to determine the extent to which the app supports secure communication processes among specialists and patients/relatives in their daily work and thus leads to a reduction in pAEs. The app helps users (skilled workers, mothers to be and relatives) to refine and improve their communication skills and, hence, to prepare for a safe birth. Controls form the data of the participants of both intervention arms of the preceding RCT study from phase 2 (historical control groups; No-Treatment CG analysis: N = 176; No-Treatment CG recruited: N = 212; Treatment CG analysis: N = 176; Treatment CG recruited: N = 212). The RCT in Phase 3 includes an intervention group who will have immediate access to the web-app after a baseline questionnaire and a waiting-list control group who will receive access to the web-app after a waiting period of 4 weeks. Recruiting is not only limited to the 2 clinics to reach a sample size with enough power to detect significant effects, but also includes a Germany-wide implementation and recruitment. This allows a first limited statement about the possible effect of a process supporting digital app. With an alpha error of 0.05 and a power of 80%, a sample of N = 352 (analysis sample) is required to be able to prove an effect of d = 0.3. Due to the historical control group, only N = 176 participants need to be analyzed for the intervention group (IG analysis). Assuming a drop-out of 20%, N = 424 participants would have to be recruited (recruitment sample). Due to the historical control group only N = 212 participants have to be recruited for the intervention group (IG recruited). The target criteria (primary: pAEs; Secondary: pAE costs, different communication models competencies, training-proximal outcomes such as outcome expectations, behavioral intention, action and coping planning, behavior, self-efficacy expectation, adherence safety culture, perceived safety culture, treatment satisfaction; covariates: sociodemographic characteristics) are evaluated statistically and clinically as in Phase 1 and 2. Group differences are checked by means of linear and general mixed models, initial values of the first measurement point are considered as covariates. Clinics are modeled as fixed effects. For the entire analysis, corresponding confidence intervals of 95 % are determined. To calculate the standardized mean difference (SMD) between the two measurement points, the non-standardized regression coefficients are standardized to the pooled standard deviation of the observed measured values. According to Cohen's recommendations, SMDs are interpreted as follows: small effect by SMD = 0.2; medium effect by SMD = 0.5; large effect by SMD = 0.8. The odds ratio of binary outcomes is subjected to a logit transformation to calculate effect strengths. To check whether the primary target criterion is moderated by external variables, reciprocal interaction terms are considered in the model estimation. Continuous moderators are standardized by z-transformation. The estimated parameter of the interaction between the z-transformed continuous variable and the effect estimator of the group difference thus represents the additional intervention effect if the potential moderator increases by one standard deviation. Participants are only included in the analysis if they participate in the corresponding follow-up survey and are analyzed according to intention to treat. Differences are interpreted as significant when the p-value of a two-sided test is <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Expectant mother or patient in gynecology and obstetrics or social support providers (spouse/partner, relative, close friend) to be recipient of the training
* Professional in a gynecology and obstetrics hospital to be trainer of the patients and the social support providers
* Aged 18 years and above
* Healthy volunteers
* Declaration of consent for participation in the study

Exclusion Criteria:

* Not proficient in the German language and/ or does not have the capability of writing
* Severe cognitive deficits (unable to read/write/answer questions) and impairments due to diagnosed brain injuries, neurological disorders, etc.
* Insufficient corrected eyesight (patients must be able to read on the cell phone)
* Participation in another research study or intervention trial conducted in the clinic
* Younger than 18 years
* High risk, emergency case
* Withdraw of consent for participation in the study at any point in time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Core competencies and preventable adverse events - specialists | 16 Months
  The core competencies of all specialists will improve measurably. Furthermore, the number of preventable adverse events (pAEs) and their associated costs should be significantly changed over time.
Core competencies surrounding communication - patients and relatives | 16 Months
  It is expected that patients/accompanying persons in the intervention group will (1) measurably improve their communication competencies with skilled employees after the intervention compared to those giving birth/accompanying persons in the control group, and (2) a higher expectation of self-efficacy in communication with skilled employees will arise. In addition, it is expected that (3) the number and severity of preventable adverse events (pAEs) in the intervention group will be measurably reduced compared to the number and severity of preventable adverse events in the control group.
Usability and effectiveness of the digital communication app | 16 Months
  The use of a digital communication app will lead to a significantly changed number, severity and cost of preventable adverse events (pAEs) in the intervention group compared to the intervention group without an app.

SECONDARY OUTCOMES:
Proximal outcomes to the online training | 16 months
  outcome expectancy, intentions, action and coping plans, behavior, self-efficacy, patient satisfaction, employee satisfaction
Covariables of the training and preventable adverse events (pAEs) | 16 months
  barriers and resources

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Lippke, Prof. Dr., Principal Investigator — Jacobs University Bremen, Germany
Locations (2):
- Germany (2):
  - Universitaetsklinikum Ulm; Klinik fuer Frauenheilkunde und Geburtshilfe, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Frankfurt; Klinik für Frauenheilkunde und Geburtshilfe, Frankfurt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pronovost PJ, Holzmueller CG, Ennen CS, Fox HE. Overview of progress in patient safety. Am J Obstet Gynecol. 2011 Jan;204(1):5-10. doi: 10.1016/j.ajog.2010.11.001. PMID 21187195
- [Background] Bartlett G, Blais R, Tamblyn R, Clermont RJ, MacGibbon B. Impact of patient communication problems on the risk of preventable adverse events in acute care settings. CMAJ. 2008 Jun 3;178(12):1555-62. doi: 10.1503/cmaj.070690. PMID 18519903
- [Background] Leonard M, Graham S, Bonacum D. The human factor: the critical importance of effective teamwork and communication in providing safe care. Qual Saf Health Care. 2004 Oct;13 Suppl 1(Suppl 1):i85-90. doi: 10.1136/qhc.13.suppl_1.i85. PMID 15465961
- [Background] Hickson GB, Clayton EW, Githens PB, Sloan FA. Factors that prompted families to file medical malpractice claims following perinatal injuries. JAMA. 1992 Mar 11;267(10):1359-63. PMID 1740858
- [Background] Olde Bekkink M, Farrell SE, Takayesu JK. Interprofessional communication in the emergency department: residents' perceptions and implications for medical education. Int J Med Educ. 2018 Oct 25;9:262-270. doi: 10.5116/ijme.5bb5.c111. PMID 30368487
- [Background] Lyndon A, Zlatnik MG, Wachter RM. Effective physician-nurse communication: a patient safety essential for labor and delivery. Am J Obstet Gynecol. 2011 Aug;205(2):91-6. doi: 10.1016/j.ajog.2011.04.021. Epub 2011 Apr 16. PMID 21640970
- [Background] Antony J, Zarin W, Pham B, Nincic V, Cardoso R, Ivory JD, Ghassemi M, Barber SL, Straus SE, Tricco AC. Patient safety initiatives in obstetrics: a rapid review. BMJ Open. 2018 Jul 6;8(7):e020170. doi: 10.1136/bmjopen-2017-020170. PMID 29982200
- [Background] Chang YS, Coxon K, Portela AG, Furuta M, Bick D. Interventions to support effective communication between maternity care staff and women in labour: A mixed-methods systematic review. Midwifery. 2018 Apr;59:4-16. doi: 10.1016/j.midw.2017.12.014. Epub 2017 Dec 27. PMID 29351865
- [Background] Hannawa AF. Disclosing medical errors to patients: effects of nonverbal involvement. Patient Educ Couns. 2014 Mar;94(3):310-3. doi: 10.1016/j.pec.2013.11.007. Epub 2013 Nov 28. PMID 24332933
- [Background] Zech A, Gross B, Jasper-Birzele C, Jeschke K, Kieber T, Lauterberg J, Lazarovici M, Pruckner S, Rall M, Reddersen S, Sandmeyer B, Scholz C, Stricker E, Urban B, Zobel A, Singer I. Evaluation of simparteam - a needs-orientated team training format for obstetrics and neonatology. J Perinat Med. 2017 Apr 1;45(3):333-341. doi: 10.1515/jpm-2016-0091. PMID 27464031
- [Background] Berg CJ, Harper MA, Atkinson SM, Bell EA, Brown HL, Hage ML, Mitra AG, Moise KJ Jr, Callaghan WM. Preventability of pregnancy-related deaths: results of a state-wide review. Obstet Gynecol. 2005 Dec;106(6):1228-34. doi: 10.1097/01.AOG.0000187894.71913.e8. PMID 16319245
- [Background] Tanaka K, Eriksson L, Asher R, Obermair A. Incidence of adverse events, preventability and mortality in gynaecological hospital admissions: A systematic review and meta-analysis. Aust N Z J Obstet Gynaecol. 2019 Apr;59(2):195-200. doi: 10.1111/ajo.12937. Epub 2019 Jan 20. PMID 30663036
- [Background] Panagioti M, Geraghty K, Johnson J, Zhou A, Panagopoulou E, Chew-Graham C, Peters D, Hodkinson A, Riley R, Esmail A. Association Between Physician Burnout and Patient Safety, Professionalism, and Patient Satisfaction: A Systematic Review and Meta-analysis. JAMA Intern Med. 2018 Oct 1;178(10):1317-1331. doi: 10.1001/jamainternmed.2018.3713. PMID 30193239 (Retraction: PMID 32421149 JAMA Intern Med. 2020 Jul 1;180(7):931)
- [Background] Welp A, Meier LL, Manser T. Emotional exhaustion and workload predict clinician-rated and objective patient safety. Front Psychol. 2015 Jan 22;5:1573. doi: 10.3389/fpsyg.2014.01573. eCollection 2014. PMID 25657627
- [Background] Welp A, Meier LL, Manser T. The interplay between teamwork, clinicians' emotional exhaustion, and clinician-rated patient safety: a longitudinal study. Crit Care. 2016 Apr 19;20(1):110. doi: 10.1186/s13054-016-1282-9. PMID 27095501
- [Background] Morony S, Weir K, Duncan G, Biggs J, Nutbeam D, Mccaffery KJ. Enhancing communication skills for telehealth: development and implementation of a Teach-Back intervention for a national maternal and child health helpline in Australia. BMC Health Serv Res. 2018 Mar 7;18(1):162. doi: 10.1186/s12913-018-2956-6. PMID 29514642
- [Background] Avula R, Menon P, Saha KK, Bhuiyan MI, Chowdhury AS, Siraj S, Haque R, Jalal CS, Afsana K, Frongillo EA. A program impact pathway analysis identifies critical steps in the implementation and utilization of a behavior change communication intervention promoting infant and child feeding practices in Bangladesh. J Nutr. 2013 Dec;143(12):2029-37. doi: 10.3945/jn.113.179085. Epub 2013 Sep 25. PMID 24068790
- [Background] Tan DJA, Sultana R, Han NLR, Sia ATH, Sng BL. Investigating determinants for patient satisfaction in women receiving epidural analgesia for labour pain: a retrospective cohort study. BMC Anesthesiol. 2018 May 9;18(1):50. doi: 10.1186/s12871-018-0514-8. PMID 29743028
- [Background] Weis J, Zoffmann V, Egerod I. Improved nurse-parent communication in neonatal intensive care unit: evaluation and adjustment of an implementation strategy. J Clin Nurs. 2014 Dec;23(23-24):3478-89. doi: 10.1111/jocn.12599. Epub 2014 Apr 3. PMID 24698260
- [Background] Bolognesi M, Nigg CR, Massarini M, Lippke S. Reducing obesity indicators through brief physical activity counseling (PACE) in Italian primary care settings. Ann Behav Med. 2006 Apr;31(2):179-85. doi: 10.1207/s15324796abm3102_10. PMID 16542133
- [Background] Omura M, Maguire J, Levett-Jones T, Stone TE. The effectiveness of assertiveness communication training programs for healthcare professionals and students: A systematic review. Int J Nurs Stud. 2017 Nov;76:120-128. doi: 10.1016/j.ijnurstu.2017.09.001. Epub 2017 Sep 5. PMID 28964979
- [Background] Haug S, Meyer C, Dymalski A, Lippke S, John U. Efficacy of a text messaging (SMS) based smoking cessation intervention for adolescents and young adults: study protocol of a cluster randomised controlled trial. BMC Public Health. 2012 Jan 19;12:51. doi: 10.1186/1471-2458-12-51. PMID 22260736
- [Background] Lippke S, Fleig L, Wiedemann AU, Schwarzer R. A Computerized Lifestyle Application to Promote Multiple Health Behaviors at the Workplace: Testing Its Behavioral and Psychological Effects. J Med Internet Res. 2015 Oct 1;17(10):e225. doi: 10.2196/jmir.4486. PMID 26429115
- [Background] Duan YP, Liang W, Guo L, Wienert J, Si GY, Lippke S. Evaluation of a Web-Based Intervention for Multiple Health Behavior Changes in Patients With Coronary Heart Disease in Home-Based Rehabilitation: Pilot Randomized Controlled Trial. J Med Internet Res. 2018 Nov 19;20(11):e12052. doi: 10.2196/12052. PMID 30455167
- [Background] Storm V, Dorenkamper J, Reinwand DA, Wienert J, De Vries H, Lippke S. Effectiveness of a Web-Based Computer-Tailored Multiple-Lifestyle Intervention for People Interested in Reducing their Cardiovascular Risk: A Randomized Controlled Trial. J Med Internet Res. 2016 Apr 11;18(4):e78. doi: 10.2196/jmir.5147. PMID 27068880
- [Background] Lippke S, Schwarzer R, Ziegelmann JP, Scholz U, Schuz B. Testing stage-specific effects of a stage-matched intervention: a randomized controlled trial targeting physical exercise and its predictors. Health Educ Behav. 2010 Aug;37(4):533-46. doi: 10.1177/1090198109359386. Epub 2010 Jun 14. PMID 20547760
- [Background] Lippke S, Plotnikoff RC. Testing two principles of the Health Action Process Approach in individuals with type 2 diabetes. Health Psychol. 2014 Jan;33(1):77-84. doi: 10.1037/a0030182. Epub 2012 Oct 22. PMID 23088172
- [Background] Lippke S, Corbet JM, Lange D, Parschau L, Schwarzer R. Intervention Engagement Moderates the Dose-Response Relationships in a Dietary Intervention. Dose Response. 2016 Mar 16;14(1):1559325816637515. doi: 10.1177/1559325816637515. eCollection 2016 Jan-Mar. PMID 27069440
- [Background] Sprangers S, Dijkstra K, Romijn-Luijten A. Communication skills training in a nursing home: effects of a brief intervention on residents and nursing aides. Clin Interv Aging. 2015 Jan 20;10:311-9. doi: 10.2147/CIA.S73053. eCollection 2015. PMID 25653513
- [Background] Zhang CQ, Zhang R, Schwarzer R, Hagger MS. A meta-analysis of the health action process approach. Health Psychol. 2019 Jul;38(7):623-637. doi: 10.1037/hea0000728. Epub 2019 Apr 11. PMID 30973747
- [Background] Reyes Fernandez B, Lippke S, Knoll N, Blanca Moya E, Schwarzer R. Promoting action control and coping planning to improve hand hygiene. BMC Public Health. 2015 Sep 25;15:964. doi: 10.1186/s12889-015-2295-z. PMID 26407591
- [Background] Lhakhang P, Lippke S, Knoll N, Schwarzer R. Evaluating brief motivational and self-regulatory hand hygiene interventions: a cross-over longitudinal design. BMC Public Health. 2015 Feb 4;15:79. doi: 10.1186/s12889-015-1453-7. PMID 25649150
- [Background] Ernsting A, Gellert P, Schneider M, Lippke S. A mediator model to predict workplace influenza vaccination behaviour--an application of the health action process approach. Psychol Health. 2013;28(5):579-92. doi: 10.1080/08870446.2012.753072. Epub 2012 Dec 24. PMID 23259583
- [Background] Alders I, Smits C, Brand P, van Dulmen S. Does patient coaching make a difference in patient-physician communication during specialist consultations? A systematic review. Patient Educ Couns. 2017 May;100(5):882-896. doi: 10.1016/j.pec.2016.12.029. Epub 2016 Dec 29. PMID 28089309
- [Background] Belkora J, Volz S, Loth M, Teng A, Zarin-Pass M, Moore D, Esserman L. Coaching patients in the use of decision and communication aids: RE-AIM evaluation of a patient support program. BMC Health Serv Res. 2015 May 28;15:209. doi: 10.1186/s12913-015-0872-6. PMID 26017564
- [Background] Dykes PC, Rozenblum R, Dalal A, Massaro A, Chang F, Clements M, Collins S, Donze J, Fagan M, Gazarian P, Hanna J, Lehmann L, Leone K, Lipsitz S, McNally K, Morrison C, Samal L, Mlaver E, Schnock K, Stade D, Williams D, Yoon C, Bates DW. Prospective Evaluation of a Multifaceted Intervention to Improve Outcomes in Intensive Care: The Promoting Respect and Ongoing Safety Through Patient Engagement Communication and Technology Study. Crit Care Med. 2017 Aug;45(8):e806-e813. doi: 10.1097/CCM.0000000000002449. PMID 28471886
- [Background] Ammentorp J, Graugaard LT, Lau ME, Andersen TP, Waidtlow K, Kofoed PE. Mandatory communication training of all employees with patient contact. Patient Educ Couns. 2014 Jun;95(3):429-32. doi: 10.1016/j.pec.2014.03.005. Epub 2014 Mar 12. PMID 24666773
- [Background] Emani SS, Allan CK, Forster T, Fisk AC, Lagrasta C, Zheleva B, Weinstock P, Thiagarajan RR. Simulation training improves team dynamics and performance in a low-resource cardiac intensive care unit. Ann Pediatr Cardiol. 2018 May-Aug;11(2):130-136. doi: 10.4103/apc.APC_117_17. PMID 29922009
- [Background] Forster AJ, Fung I, Caughey S, Oppenheimer L, Beach C, Shojania KG, van Walraven C. Adverse events detected by clinical surveillance on an obstetric service. Obstet Gynecol. 2006 Nov;108(5):1073-83. doi: 10.1097/01.AOG.0000242565.28432.7c. PMID 17077227
- [Background] Pettker CM. Systematic approaches to adverse events in obstetrics, Part I: Event identification and classification. Semin Perinatol. 2017 Apr;41(3):151-155. doi: 10.1053/j.semperi.2017.03.003. Epub 2017 May 23. PMID 28549789
- [Background] Ellenbecker CH, Byleckie JJ. Home Healthcare Nurses' Job Satisfaction Scale: refinement and psychometric testing. J Adv Nurs. 2005 Oct;52(1):70-8. doi: 10.1111/j.1365-2648.2005.03556.x. PMID 16149983
- [Background] Bussing A, Perrar KM. [Burnout measurement. Study of a German version of the Maslach Burnout Inventory (MBI-D)]. Pflege Z. 1994 Mar;47(3):suppl 20-30. No abstract available. German. PMID 8004334
- [Background] Stevenson RJ, Case TI, Hodgson D, Porzig-Drummond R, Barouei J, Oaten MJ. A scale for measuring hygiene behavior: development, reliability and validity. Am J Infect Control. 2009 Sep;37(7):557-64. doi: 10.1016/j.ajic.2009.01.003. Epub 2009 Apr 10. PMID 19362392
- [Background] Hellings J, Schrooten W, Klazinga N, Vleugels A. Challenging patient safety culture: survey results. Int J Health Care Qual Assur. 2007;20(7):620-32. doi: 10.1108/09526860710822752. PMID 18030963
- [Background] Nabhan A, Ahmed-Tawfik MS. Understanding and attitudes towards patient safety concepts in obstetrics. Int J Gynaecol Obstet. 2007 Sep;98(3):212-6. doi: 10.1016/j.ijgo.2007.05.012. Epub 2007 Jul 5. PMID 17618630
- [Background] Whittal A, Lippke S. Investigating patients with an immigration background in Canada: relationships between individual immigrant attitudes, the doctor-patient relationship, and health outcomes. BMC Public Health. 2016 Jan 12;16:23. doi: 10.1186/s12889-016-2695-8. PMID 26753690
- [Background] Whittal A, Hanke K, Lippke S. Investigating acculturation orientations of patients with an immigration background and doctors in Canada: implications for medical advice adherence. Qual Life Res. 2017 May;26(5):1223-1232. doi: 10.1007/s11136-016-1438-8. Epub 2016 Oct 19. PMID 27761682
- [Background] Hannawa AF, Roter DL. TRACEing the roots: a diagnostic "Tool for Retrospective Analysis of Critical Events". Patient Educ Couns. 2013 Nov;93(2):230-8. doi: 10.1016/j.pec.2013.06.019. Epub 2013 Jul 23. PMID 23891421
- [Background] Teunissen E, Gravenhorst K, Dowrick C, Van Weel-Baumgarten E, Van den Driessen Mareeuw F, de Brun T, Burns N, Lionis C, Mair FS, O'Donnell C, O'Reilly-de Brun M, Papadakaki M, Saridaki A, Spiegel W, Van Weel C, Van den Muijsenbergh M, MacFarlane A. Implementing guidelines and training initiatives to improve cross-cultural communication in primary care consultations: a qualitative participatory European study. Int J Equity Health. 2017 Feb 10;16(1):32. doi: 10.1186/s12939-017-0525-y. PMID 28222736
- [Background] Meeks DW, Smith MW, Taylor L, Sittig DF, Scott JM, Singh H. An analysis of electronic health record-related patient safety concerns. J Am Med Inform Assoc. 2014 Nov-Dec;21(6):1053-9. doi: 10.1136/amiajnl-2013-002578. Epub 2014 Jun 20. PMID 24951796
- [Background] van Dinter-Douma EE, de Vries NE, Aarts-Greven M, Stramrood CAI, van Pampus MG. Screening for trauma and anxiety recognition: knowledge, management and attitudes amongst gynecologists regarding women with fear of childbirth and postpartum posttraumatic stress disorder. J Matern Fetal Neonatal Med. 2020 Aug;33(16):2759-2767. doi: 10.1080/14767058.2018.1560409. Epub 2019 Jan 4. PMID 30563384
- [Background] Taylor LJ, Adkins S, Hoel AW, Hauser J, Suwanabol P, Wood G, Anderson W, Branson C, Skube S, Johnson SK, Zelenski A, Tucholka JL, Campbell TC, Schwarze ML. Using Implementation Science to Adapt a Training Program to Assist Surgeons with High-Stakes Communication. J Surg Educ. 2019 Jan-Feb;76(1):165-173. doi: 10.1016/j.jsurg.2018.05.015. Epub 2018 Jul 4. PMID 30626527
- [Background] Karger A, Geiser F, Vitinius F, Sonntag B, Schultheis U, Hey B, Radbruch L, Ernstmann N, Petermann-Meyer A. Communication Skills Trainings: Subjective Appraisal of Physicians from Five Cancer Centres in North Rhine, Germany. Oncol Res Treat. 2017;40(9):496-501. doi: 10.1159/000479113. Epub 2017 Jul 28. PMID 28750399
- [Background] Yu L, Kronen RJ, Simon LE, Stoll CRT, Colditz GA, Tuuli MG. Prophylactic negative-pressure wound therapy after cesarean is associated with reduced risk of surgical site infection: a systematic review and meta-analysis. Am J Obstet Gynecol. 2018 Feb;218(2):200-210.e1. doi: 10.1016/j.ajog.2017.09.017. Epub 2017 Sep 23. PMID 28951263
- [Background] Nigam A, Huising R, Golden BR. Improving hospital efficiency: a process model of organizational change commitments. Med Care Res Rev. 2014 Feb;71(1):21-42. doi: 10.1177/1077558713504464. Epub 2013 Oct 16. PMID 24132582
- [Background] Bashour HN, Kanaan M, Kharouf MH, Abdulsalam AA, Tabbaa MA, Cheikha SA. The effect of training doctors in communication skills on women's satisfaction with doctor-woman relationship during labour and delivery: a stepped wedge cluster randomised trial in Damascus. BMJ Open. 2013 Aug 14;3(8):e002674. doi: 10.1136/bmjopen-2013-002674. PMID 23945729
- [Background] Crofts JF, Bartlett C, Ellis D, Winter C, Donald F, Hunt LP, Draycott TJ. Patient-actor perception of care: a comparison of obstetric emergency training using manikins and patient-actors. Qual Saf Health Care. 2008 Feb;17(1):20-4. doi: 10.1136/qshc.2006.021873. PMID 18245215
- [Background] Schrappe M. APS-Weißbuch Patientensicherheit. Sicherheit in der Gesundheitsversorgung: neu denken, gezielt verbessern [APS Report on Patient safety]. 1st ed. Berlin: Medizinisch Wissenschaftliche Verlagsgesellschaft; 2018.
- [Background] Lippke S, Wienert J, Keller FM, Derksen C, Welp A, Kotting L, Hofreuter-Gatgens K, Muller H, Louwen F, Weigand M, Ernst K, Kraft K, Reister F, Polasik A, Huener Nee Seemann B, Jennewein L, Scholz C, Hannawa A. Communication and patient safety in gynecology and obstetrics - study protocol of an intervention study. BMC Health Serv Res. 2019 Nov 28;19(1):908. doi: 10.1186/s12913-019-4579-y. PMID 31779620
- [Result] Derksen C, Keller FM, Lippke S. Obstetric Healthcare Workers' Adherence to Hand Hygiene Recommendations during the COVID-19 Pandemic: Observations and Social-Cognitive Determinants. Appl Psychol Health Well Being. 2020 Dec;12(4):1286-1305. doi: 10.1111/aphw.12240. Epub 2020 Oct 5. PMID 33016518
- [Result] Schmiedhofer M, Derksen C, Keller FM, Dietl JE, Haussler F, Strametz R, Koester-Steinebach I, Lippke S. Barriers and Facilitators of Safe Communication in Obstetrics: Results from Qualitative Interviews with Physicians, Midwives and Nurses. Int J Environ Res Public Health. 2021 Jan 21;18(3):915. doi: 10.3390/ijerph18030915. PMID 33494448
- [Result] Keller, F., Derksen, C., Schmiedhofer, M., Welp, A., Kötting, L. and Lippke, S., 2020. Patientensicherheit und wahrgenommene Risiken für Vermeidbare Unerwünschte Ereignisse aus Sicht von Patienten und Beschäftigten im Gesundheitswesen. Monitor Versorgungsforschung, 13(05/2020), pp.83-89. doi:http://doi.org/10.24945/MVF.05.20.1866-0533.2251
- [Result] Derksen C, Kotting L, Keller FM, Schmiedhofer M, Lippke S. Psychological Intervention to Improve Communication and Patient Safety in Obstetrics: Examination of the Health Action Process Approach. Front Psychol. 2022 Feb 18;13:771626. doi: 10.3389/fpsyg.2022.771626. eCollection 2022. PMID 35250715
- [Result] Huner B, Derksen C, Schmiedhofer M, Lippke S, Janni W, Scholz C. Preventable Adverse Events in Obstetrics-Systemic Assessment of Their Incidence and Linked Risk Factors. Healthcare (Basel). 2022 Jan 4;10(1):97. doi: 10.3390/healthcare10010097. PMID 35052261
- [Result] Keller FM, Derksen C, Kotting L, Schmiedhofer M, Lippke S. Development of the perceptions of preventable adverse events assessment tool (PPAEAT): measurement properties and patients' mental health status. Int J Qual Health Care. 2021 Apr 16;33(2):mzab063. doi: 10.1093/intqhc/mzab063. PMID 33822086
- [Result] Lippke S, Derksen C, Keller FM, Kotting L, Schmiedhofer M, Welp A. Effectiveness of Communication Interventions in Obstetrics-A Systematic Review. Int J Environ Res Public Health. 2021 Mar 5;18(5):2616. doi: 10.3390/ijerph18052616. PMID 33807819
- [Result] Schmiedhofer M, Derksen C, Dietl JE, Haussler F, Louwen F, Huner B, Reister F, Strametz R, Lippke S. Birthing under the Condition of the COVID-19 Pandemic in Germany: Interviews with Mothers, Partners, and Obstetric Health Care Workers. Int J Environ Res Public Health. 2022 Jan 28;19(3):1486. doi: 10.3390/ijerph19031486. PMID 35162509
- [Derived] Kotting L, Anand-Kumar V, Keller FM, Henschel NT, Lippke S. Effective Communication Supported by an App for Pregnant Women: Quantitative Longitudinal Study. JMIR Hum Factors. 2024 Apr 26;11:e48218. doi: 10.2196/48218. PMID 38669073
- [Derived] Kotting L, Derksen C, Keller FM, Lippke S. Comparing the Effectiveness of a Web-Based Application With a Digital Live Seminar to Improve Safe Communication for Pregnant Women: 3-Group Partially Randomized Controlled Trial. JMIR Pediatr Parent. 2023 Jul 24;6:e44701. doi: 10.2196/44701. PMID 37486755
- [Derived] Huner B, Derksen C, Schmiedhofer M, Lippke S, Riedmuller S, Janni W, Reister F, Scholz C. Reducing preventable adverse events in obstetrics by improving interprofessional communication skills - Results of an intervention study. BMC Pregnancy Childbirth. 2023 Jan 23;23(1):55. doi: 10.1186/s12884-022-05304-8. PMID 36690974
- [Derived] Derksen C, Dietl JE, Haeussler FE, Steinherr Zazo M, Schmiedhofer M, Lippke S. Behavior change training for pregnant women's communication during birth: A randomized controlled trial. Appl Psychol Health Well Being. 2023 Aug;15(3):865-883. doi: 10.1111/aphw.12413. Epub 2022 Nov 15. PMID 36380576
- [Derived] Keller FM, Dahmen A, Derksen C, Kotting L, Lippke S. Psychosomatic Rehabilitation Patients and the General Population During COVID-19: Online Cross-sectional and Longitudinal Study of Digital Trainings and Rehabilitation Effects. JMIR Ment Health. 2021 Aug 26;8(8):e30610. doi: 10.2196/30610. PMID 34270444
- See also: Project description and outline of partners — https://www.jacobs-university.de/teambaby

DOCUMENTS (1):
  • Study Protocol (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT03855735/Prot_000.pdf